CLINICAL TRIAL: NCT04362839
Title: A Phase I Clinical Trial of Regorafenib, Nivolumab, and Ipilimumab in Advanced Chemotherapy Resistant Metastatic MSS Colorectal Cancer
Brief Title: Regorafenib, Ipilimumab and Nivolumab for the Treatment of Chemotherapy Resistant Microsatellite Stable Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19417; NCI-2020-01818 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19417 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Colon Adenocarcinoma; Metastatic Colon Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (regorafenib, nivolumab, ipilimumab) (Experimental): Patients receive regorafenib PO QD on days 1-21, nivolumab IV over 30 minutes Q2W, and ipilimumab IV over 30 minutes Q6W. Cycles repeat every 28 day for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Regorafenib

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga

SUMMARY:
This phase I trial studies the side effects and best dose of regorafenib when given together with ipilimumab and nivolumab in treating patients with microsatellite stable colorectal cancer that has spread to other places in the body (metastatic) and remains despite chemotherapy treatment (resistant). Regorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving regorafenib, ipilimumab and nivolumab may slow the tumor growth and/or shrink the tumor size in patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended dose level of the combination of regorafenib, nivolumab and ipilimumab in patients with advanced metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. Assess the objective overall response rate per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

II. Estimate the duration of response, duration of stable disease (SD), progression free survival (PFS), and overall survival (OS).

III. Describe the safety of this regimen as determined by frequency and severity of associated adverse events.

EXPLORATORY OBJECTIVES:

I. Correlate the presence of colony stimulating factor 1 receptor (CSF1R)+ macrophages, regulatory T cells (Tregs), TILs (tumor infiltrating lymphocytes) and tumor PD-L1, CTLA-4 and PD1 expression (at baseline and post treatment) on tumor biopsies with response rate.

II. Characterize the systemic immune alteration through evaluation of mandatory pre and post cycle 1, and cycle 2, and at progression blood draws.

OUTLINE: This is a dose-escalation study of regorafenib.

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21, nivolumab intravenously (IV) over 30 minutes every 2 weeks (Q2W), and ipilimumab IV over 30 minutes every 6 weeks (Q6W). Cycles repeat every 28 day for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent must be obtained prior to conducting any study-specific procedures
* Histological or cytological confirmed advanced, metastatic, or progressive mismatch repair protein proficient (pMMR)/microsatellite stable (MSS) adenocarcinoma of colon or rectum

  * Microsatellite status should be performed per local standard of practice (e.g., immunohistochemistry [IHC] and/or polymerase chain reaction [PCR], or next-generation sequencing). Only participants with pMMR/MSS metastatic colorectal cancer (mCRC) are eligible
* Known extended RAS and BRAF status as per local standard of practice
* Participant must have progressed following exposure of all the following agents or below:

  * Prior exposure to the following:

    * Fluoropyrimidines (capecitabine or fluorouracil [5-FU])
    * Irinotecan
    * Oxaliplatin
    * Anti-EGFR therapy if RAS and BRAF wild type with left colon primary
  * Patient must have evidence of progression on or after the last treatment regimen received and within 6 months prior to study enrollment
  * Patients who were intolerant to prior systemic chemotherapy regimens are eligible if there is documented evidence of clinically significant intolerance despite adequate supportive measures
  * Adjuvant/neoadjuvant chemotherapy can be considered as one line of chemotherapy for advanced/metastatic disease if the participant had disease recurrence within 6 months of completion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Total bilirubin =< 1.5 x the upper limit of normal (ULN) (performed within 7 days before treatment initiation)
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN if no liver metastases; ALT or AST =< 5 x ULN allowed for patients with liver involvement (performed within 7 days before treatment initiation)
* Platelet count >= 100,000 /mm^3 (performed within 7 days before treatment initiation)
* Hemoglobin (Hb) >= 9 g/dL (performed within 7 days before treatment initiation)
* White blood cells (WBC) >= 2000/uL (performed within 7 days before treatment initiation)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (performed within 7 days before treatment initiation)
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 40 mL/min (measured or calculated using the Cockcroft-Gault formula) (performed within 7 days before treatment initiation)
* Measurable disease as determined by RECISTv1.1
* Provision of recent tumor tissue (as defined below) is mandatory for all participants at screening (Formalin-fixed paraffin-embedded block or minimum of 20 slides)

  * Tumor tissue obtained within 180 days of enrollment and after the last dose of most recent anti-cancer therapy
  * Or a new biopsy Exceptions for patients with no recent baseline tumor tissues or biopsies may be considered after documented discussion and approval with the principal investigator (PI) of the study
* Anticipated life expectancy greater than 3 months
* Be able to swallow and absorb oral tablets
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study intervention and 120 days after last dose of regorafenib and 5 months after the last dose of nivolumab. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study intervention and 120 days after last dose of regorafenib and 7 months after the last dose of nivolumab. In addition, male participants must be willing to refrain from sperm donation during this time. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Participants with microsatellite instability high (MSI-H) colorectal cancer
* Prior therapy with regorafenib, anti-PD-1, PD-L1, or CTLA-4 inhibitors
* Systemic anti-cancer treatment within 14 days or less than 5 half-lives (whichever is shorter) of the first dose of study treatment
* Has unresolved clinically significant toxicity of greater than or equal to National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) (NCI-CTCAE, v5.0) grade 2 attributed to any prior therapies (excluding anemia, lymphopenia, alopecia, skin pigmentation, and platinum-induced neurotoxicity)
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
* Congestive heart failure >= New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), myocardial infarction less than 6 months before start of study drug
* Uncontrolled cardiac arrhythmias
* Poorly controlled hypertension, defined as a blood pressure consistently above 150/90 mmHg despite optimal medical management
* Persistent proteinuria of NCI-CTCAE grade 3. Urine dipstick result of 3+ or abnormal, based on type of urine test strip used, is allowed if protein excretion (estimated by urine protein/creatinine ratio on a random urine sample) is < 3.5 g/24 hr
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Non-healing wound, non-healing ulcer, or non-healing bone fracture
* Participants with evidence or history of any bleeding diathesis, irrespective of severity
* Any hemorrhage or bleeding event >= NCI-CTCAE grade 3 within 28 days prior to the start of study medication
* Significant acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or >= NCI-CTCAE grade 2 diarrhea of any etiology
* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus (T1DM), hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* History of interstitial lung disease
* Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission prior to study entry and no additional therapy is required or anticipated to be required during the study period
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy
* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed treatment (such as radiotherapy or surgery). Participants with stable CNS disease or previously treated lesions are eligible for study entry. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of 10 mg daily prednisone (or equivalent)
* Ongoing infection > grade 2 NCI-CTCAE requiring systemic therapy
* Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies)
* Any positive test result for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating presence of virus, e.g. hepatitis B surface antigen (HBsAg, Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive (except if HCV-ribonucleic acid [RNA] negative)
* Pregnancy or breast feeding
* Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up (FU) schedule
* Previous treatment with live vaccine within 30 days of planned start of study drugs (seasonal flu vaccines that do not contain a live virus are permitted)
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Recommended dose level of the combination | Up to 90 days post treatment
  Toxicities will be graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v). 5.0. Dose limiting toxicity (DLT) will be graded per CTCAE v5.0. Any of the following adverse events occurring during the primary DLT observation period (4 weeks, from the time of first administration of regorafenib, ipilimumab and nivolumab[cycle 1 day 1] until the planned administration of the second cycle of regorafenib (cycle 2 day 1) that are at least probable attributable to many of the 3 agents or their combination will be classified as a DLT.

SECONDARY OUTCOMES:
Progression-free survival | Time to disease progression/ relapse or death as a result of any cause, assessed up to 5 years
  Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. Will be summarized using the Kaplan-Meier method.
Duration of response | Time to progression or death, assessed up to 5 years
  Assessed using RECIST v 1.1. Duration of response (possibly censored) will be reported for each response.
Overall survival | Time to death as a result of any cause, assessed up to 5 years
  Assessed using RECIST v 1.1. Will be summarized using the Kaplan-Meier method.
Objective response rate (ORR) | Up to 5 years post treatment
  ORR is defined as the percentage of measurable disease participants who have achieved either complete response (CR) or partial response (PR). Assessed using RECIST v 1.1.

OTHER OUTCOMES:
Immune response | Baseline, assessed up to 5 years post treatment
  Correlative studies using serial tumor tissue and blood samples will assess immune response at pre-treatment and post-treatment. Will be summarized using exploratory methods. Changes in tumor and blood measurements from pre-treatment to post-treatment will be displayed graphically and summarized with responding individuals identified. Academic standard statistical methods will be used for these exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Fakih M, Sandhu J, Lim D, Li X, Li S, Wang C. Regorafenib, Ipilimumab, and Nivolumab for Patients With Microsatellite Stable Colorectal Cancer and Disease Progression With Prior Chemotherapy: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):627-634. doi: 10.1001/jamaoncol.2022.7845. PMID 36892833